CLINICAL TRIAL: NCT05665920
Title: Clinical Trial to Assess the Efficacy and Safety of Ultra_HYPofractionated RadiotHerapy in Women With BrEast CaNcer Receiving Regional Nodal Radiation vs Nodal Moderate Hypofractionated Radiotherapy
Brief Title: Efficacy and Safety of Ultra_HYPofractionated RadiotHerapy in Women With BrEast CaNcer Receiving Regional Nodal Radiation vs Nodal Moderate Hypofractionated Radiotherapy
Acronym: HYPHEN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Brasileiro de Controle do Cancer (Other)
Responsible Party: Principal Investigator, Eduardo Barbieri, Principal Investigator, Instituto Brasileiro de Controle do Cancer
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 60905722.0.0000.0072
Record Dates: First submitted 2022-12-16; First posted 2022-12-27 (Actual); Last update posted 2022-12-29 (Actual); Status verified 2022-12

CONDITIONS: Malignant Breast Neoplasm
Keywords: Dose splitting; Acute and late toxicity; Locoregional drainage irradiation; Breast neoplasm; Overall survival; Disease-free survival; Locoregional control
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Whole breast Radiotherapy (Active Comparator): Standard Radiation: Whole Breast Irradiation, at 40 Gy, in 15 fractions and drainage
  Interventions: Radiation: Standard Radiation
- Ultra-hypofractionated whole breast radiotherapy (Experimental): Ultra-hypofractionated radiation: Ultra-hypofractionated whole breast radiotherapy, 26 Gray (26Gy) in 5 fractions for one week
  Interventions: Radiation: Ultra-hypofractionated whole breast radiotherapy

INTERVENTIONS:
Radiation: Ultra-hypofractionated whole breast radiotherapy — Ultra-hypofractionated whole breast radiotherapy, 26 Gray (26Gy) in 5 fractions for one week
  Arms: Ultra-hypofractionated whole breast radiotherapy
Radiation: Standard Radiation — Standard Radiation: Whole Breast Irradiation, at 40 Gy, in 15 fractions and drainage
  Arms: Standard Whole breast Radiotherapy

SUMMARY:
The reduction in the number of fractions in radiotherapy is especially attractive in several senses, and even more so considering breast cancer, which has a high incidence and generally favorable prognosis. Thus, as a reference Institution, the investigators intend to start the treatment of selected patients with a radiotherapy scheme of 26 Gy / 5 fractions in one week, in a controlled manner, through this project.The investigators consider the moment extremely propitious to start the study, as in addition to having the first publication of a large randomized study, proving the effectiveness and safety of the strategy, the investigators will be able to benefit more patients and the health system itself by minimizing the daily visits of these patients at the hospital.

DETAILED DESCRIPTION:
This is a prospective, interventional, exploratory, controlled, randomized study in a 1:1 ratio, to be carried out in a single center, and seeks to evaluate the safety and efficacy of hypofractionated irradiation in women with breast cancer who receive nodal irradiation regional.

ELIGIBILITY:
Inclusion Criteria:

* Information to the patient and signed informed consent;
* Women aged ≥18 years;
* Breast conserving surgery;
* Invasive adenocarcinoma (except classic invasive lobular carcinoma);
* TNM (Tumor, Nodes, Metastasis) pathologic stage pT1-3 and pN1-3a M0, with indication of lymphatic drainage according to institutional protocol;
* Eastern Cooperative Oncology Group (ECOG) 0 -1;
* Minimum microscopic margin of non-cancerous tissue of 2 mm (excluding deep margin if in the deep fascia);
* No previous breast or mediastinal radiotherapy;
* No hematogenous metastases;
* Ability to carry out long-term follow-up;

Exclusion Criteria:

* Previous local irradiation;
* Concomitant chemotherapy. Concomitance with trastuzumab or hormone blockade will be allowed;
* Histology of metaplastic carcinoma;
* History of another neoplasm: non-melanoma skin cancer, carcinoma in situ of the uterine cervix. Another neoplasm treated with curative intent and without evidence of disease in the last 5 years will be allowed.
* Diagnosis of autoimmune and connective tissue diseases;
* Diagnosis of genetic alterations in cell repair genes (Ex: Fanconi anemia, ataxia teleangiectasia);
* Indication of internal breast irradiation.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2022-10-18 (Actual); Primary Completion 2027-10-18 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Locoregional recurrence (LRR) | 10 years
  To estimate and compare the rate of local recurrence between the experimental and control arms.

SECONDARY OUTCOMES:
Overall survival | 10 years
  Overall survival time, defined as number of days from date of initial diagnosis until death or end of follow-up.
Disease-free survival | 10 years
  Disease-free survival, defined as number of days from surgery until the first occurrence of local recurrence, distant metastases, tumor-related death, death without prior progression, or end of follow-up.
Locoregional control | 10 years
  Locoregional control defined as biopsy-proven recurrence of breast cancer involving the chest wall, breast, axilla, internal breast or supraclavicular nodes.
Early and late adverse effects in normal tissues | 10 years
  To evaluate the results reported by patient and evaluated by doctors, as well as, photographic assessments.
Late adverse effects | 10 years
  To evaluate if the patient had symptoms of swelling or edema in the arm, breast shrinkage, hardness, pigmentation, necrosis, pain and tenderness in the breast.
Acute toxicity rate | 10 years
  To evaluate acute toxicity rate. The maximum grade for acute toxicity will be recorded for each patient at each treatment evaluation using RTOG (Radiation Therapy Oncology Group).
Evaluation of quality of life change by European Organization for Research and Treatment of Cancer Breast-Cancer-Specific Quality of Life Questionnaire (EORTC QLQ-BR23) | Baseline and 3 months, 6 months, 12 months, 2 years, 10 years after treatment end
  To evaluate the patient quality of life with the help of the European Organization for Research and Treatment of Cancer Breast-Cancer-Specific Quality of Life Questionnaire (EORTC QLQ-BR23). The 23-item EORTC QLQ BR23 contains two breast cancer specific functional scales (body image and sexuality) and three symptom scales evaluating arm symptoms, breast symptoms, and systemic therapy symptoms. The minimum and maximum values are 0 and 100, and higher scores mean a better outcome.
Measurement Satisfaction of Body Image of the participants | Baseline and 3 months, 6 months, 12 months after radiotherapy and 2 years, 10 years after treatment end
  To evaluate the patient quality of life and patient satisfaction with the help of the Body Image Scale (BIS). Scores are interpreted according to the guidelines of the Scoring Manual. The Body Image Scale (BIS) is a self-assessment scale designed to assess cancer patients' perceptions of their appearance and identify any changes to those perceptions resulting from a disease or a treatment. The total score ranges from 0 to 30. A higher score means a higher level of body image disturbance.

CONTACTS AND LOCATIONS:
Overall Officials: Eduardo Barbieri, Principal Investigator — IBCC Oncologia
Locations (1):
- IBCC Oncologia, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No